CLINICAL TRIAL: NCT01637688
Title: Growth and Plasma Amino Acid Levels in Infants With Cow's Milk Protein Allergy and Treated With a Newly Innovated Amino Acid Formula (NAAF) Compared to a Commercial Amino Acid Formula (AAF)
Brief Title: Growth and Plasma Amino Acids in Infants With CMPA and Treated With a Newly Innovated Amino Acid Formula
Acronym: CMPA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si262/2012
Record Dates: First submitted 2012-06-26; First posted 2012-07-11 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cow Milk Allergy
Keywords: cow milk allergy; amino acid formula
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Neocate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Amino acid formula: Comparison of growth between subjects who are fed with a newly innovated amino acid formula (NAAF) and who are fed with either Neocate or nutramigen AA.
  Interventions: Dietary Supplement: Comparison of treatment with different amino acid formulas

INTERVENTIONS:
Dietary Supplement: Comparison of treatment with different amino acid formulas — Growth and amino acid status of a newly innovated amino acid formula (NAAF) and a commercial amino acid formula (AAF)
  Other Names: Neocate; Nutramigen AA; a newly innovated amino acid formula

SUMMARY:
The purpose of this study is to determine growth and protein status of infants with cow's milk protein allergy and treated with a newly innovated amino acid formula compared to those with a commercial amino acid formula.

DETAILED DESCRIPTION:
Severe cases of cow's milk protein allergy are treated with the amino acid formula. The amino acid formula is composed of essential and non-essential amino acids, vegetable oils with or without MCT oil, and glucose polymer from various carbohydrate sources. Such formula is also fortified by minerals, trace elements,and vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Singleton
* Clinical diagnosis of cow's milk protein allergy

Exclusion Criteria:

* Other diseases

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * population who are diagnosed cow's milk protein allergy via a double-blind placebo-controlled food challenge and consume either a newly innovated amino acid formula or a commercial amino acid formula
  * population from a well-baby clinic
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Growth and protein status | 4 weeks
  * compare body weight, length, head circumference, triceps skin fold thickness, mid-arm circumference, and arm muscle area between NAAF and AAF groups
  * compare plasma amino acids, serum albumin, blood urea nitrogen, and creatinine between NAAF and AAF groups

SECONDARY OUTCOMES:
Growth | 4 weeks
  * compare weight, length, head circumference, triceps skin fold thickness, mid-arm circumference, and arm muscle area between either NAAF group or AAF group and normal infants fed with either breast milk or infant formula.
  * compare plasma amino acids between either NAAF group or AAF group and normal published data

CONTACTS AND LOCATIONS:
Overall Officials: Narumon Densupsoontorn, MD, Principal Investigator — Asso.Prof. Narumon Densupsoontorn
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Svasti J, Wasant P, Tiensuwan M, Sawangareetrakul P, Srisomsap C, Pangkanon S, Boonpuan K, Liammongkolkul S. Normal plasma free amino acid levels in Thai children. J Med Assoc Thai. 2001 Nov;84(11):1558-68. PMID 11853298
- [Result] Burks W, Jones SM, Berseth CL, Harris C, Sampson HA, Scalabrin DM. Hypoallergenicity and effects on growth and tolerance of a new amino acid-based formula with docosahexaenoic acid and arachidonic acid. J Pediatr. 2008 Aug;153(2):266-71. doi: 10.1016/j.jpeds.2008.02.043. Epub 2008 Apr 9. PMID 18534230
- See also: Educational institute web page — http://www.si.mahidol.ac.th